CLINICAL TRIAL: NCT02948478
Title: Breast Cancer and Precariousness: Influence of Socio-demographic Inequalities in Cancer Stage at Diagnosis, Treatment Management and Rehabilitation in the Ile de France Area
Brief Title: Economic and Social Disparities and Breast Cancer
Acronym: DESSEIN
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: National Cancer Institute, France (Other Government); Paris West University Nanterre La Défense (Other); Paris 12 Val de Marne University (Other); Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: K160202; ID RCB 2016-A00589-42 (Other: Agence Nationale de Sécurité du Médicament et des Produits de Santé)
Record Dates: First submitted 2016-10-26; First posted 2016-10-28 (Estimated); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Breast Cancer
Keywords: precariousness; care pathways
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Precarious patients: Precarious patients - exposed - will be those identified as precarious by at least one of the three scores (EPICES, Pascal, European Deprivation Index)
  Interventions: Other: Exposed
- Non precarious patients: Non precarious patient - non exposed - will be all the patients identified as non-precarious by the three scores (EPICES, Pascal, European Deprivation Index)
  Interventions: Other: Non exposed

INTERVENTIONS:
Other: Exposed — Precarious patients
  Groups: Precarious patients
Other: Non exposed — Non precarious patients
  Groups: Non precarious patients

SUMMARY:
Precariousness is a multifactorial concept that can be broken down in the form of economic insecurity, and / or social insecurity and / or territorial insecurity. Precariousness has an impact on health that is difficult to assess precisely because it also impacts on other factors that may themselves influence health. Therefore, the understanding of the impact of precariousness on health involves studying individuals in their context.

Our study is designed to assess the impact of precariousness on the history of breast cancer, on care pathways, on treatment and rehabilitation in a multidisciplinary contextual analysis. Indeed, the socio -economic and geographical inequalities affect the history of breast cancer, treatment and its delay and post- treatment rehabilitation.

The main objective of this project is to compare the stage of disease at diagnosis (according to the TNM classification) in deprived and non deprived patients. The secondary objectives are to compare in the two groups - the socio-economic and geographical inequalities - the direct and indirect costs related to the management, the out-of pocket costs and to describe, based on individual inequalities identified, the pathway of care of the patient.

These objectives will be pursued in the framework of an observational cohort study, prospective, multicenter (Ile de France) comparative exposed / unexposed category. Each precarious patient will be matched to a non- precarious patient in the same age group, regardless of the center. The study will include any patient resident in Ile de France seeking treatment for breast cancer, regardless of the stage.

DETAILED DESCRIPTION:
All patients seeking treatment for breast cancer, regardless of the stage, can be included in the study. Three scores of precariousness will be applied to all patients (EPICES score, Pascal score and the European Deprivation Index). Patients identified as precarious by at least one of those three scales will be in the exposed group. The others will be in the non-exposed group.

Baseline assessment T0:

Are required only the clinical examination and radiological evaluation with the tumor size and node involvement according to TNM classification. A questionnaire will be distributed including EPICES score, Pascal score and European Deprivation Index. The baseline questionnaire will also assess the socio-economic characteristics of patients and the care trajectory before arriving in the center (see appendix).

Follow-up visits:

The following questionnaire will be distributed during a consultation that is scheduled in the routine care. There will be no additional consultation imposed on the patient.

* T1: questionnaire at 3 months after inclusion
* T2: questionnaire at 6 months after inclusion
* T3: questionnaire at 12 months after inclusion

Questionnaires will be focused on direct-costs and out-of-pocket costs, socio-economical characteristics, rehabilitation, return to work.

ELIGIBILITY:
Inclusion Criteria:

- Patients ? 18 years old having a breast cancer histologically proved

Exclusion Criteria:

- Patients with a history of cancer treated in the previous five years, or with another associated untreated cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from Ile de France area having a breast cancer histologically proved and seeking for treatment. Any patient consulting for the first time in a specialized center for the treatment of breast cancer in Ile de France, whatever the stage of the disease, may potentially be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 936 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2021-02-23 (Actual); Study Completion 2021-02-23 (Actual)

PRIMARY OUTCOMES:
TNM stage | Baseline
  TNM classification according to initial clinical and radiological assessment

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte NGO, MD, Principal Investigator — AP - HP, Hôpital Européen Georges-Pompidou, Paris, France
Locations (24):
- France (24):
  - Centre Hopitalier Victor Dupouy Argenteuil, Argenteuil
  - Hôpital Jean Verdier, Bondy
  - Centre Hospitalier de Pontoise, Cergy-Pontoise
  - Hopital Privé Paule Egine, Champigny-sur-Marne
  - CH Sud Francilien, Corbeil-Essonnes
  - Centre Hospitalier Intercommunal Créteil, Créteil
  - Hôpital Henri Mondor, Créteil
  - Clinique Claude Bernard, Ermont
  - CH de Lagny sur Marne, Lagny-sur-Marne
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Institut de Cancérologie Hartmann, Levallois-Perret
  - Institut Curie Hôpital de Paris, Paris
  - Hôpital Lariboisière, Paris
  - Hôpital Saint-Louis, Paris
  - Hôpital Privé des Peupliers, Paris
  - HEGP, Paris
  - Hôpital Tenon, Paris
  - Groupe Hospitalier Paris Saint-Joseph, Paris
  - Centre Hospitalier Intercommunal Poissy Saint Germain en Laye, Poissy
  - Institut Curie Hôpital René-Huguenin site Saint-Cloud, Saint-Cloud
  - Centre Hospitalier Delafontaine, Saint-Denis
  - Institut de cancérologie Paris Nord, Sarcelles
  - Clinique de l'Estrée, Stains
  - Centre Hospitalier de Versailles, Versailles

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ngo C, Dinut A, Bochaton A, Charreire H, Despres C, Baffert S, Lecuru F, Chatellier G. From prospective clinical trial to reducing social inequalities in health: The DESSEIN trial, concept and design of a multidisciplinary study in precarious patients with breast cancer. BMC Public Health. 2019 Nov 4;19(1):1450. doi: 10.1186/s12889-019-7611-6. PMID 31684919